CLINICAL TRIAL: NCT03345433
Title: Does Interactive Group Drumming (IGD) Improve the Hospital Experience of Patients Undergoing Hematopoietic Stem Cell Transplant? - A Pilot Study
Brief Title: Interactive Group Drumming (IGD) in Hospital Experience of Patients Undergoing Hematopoietic Stem Cell Transplant - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00046180; CCCWFU 04417 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2017-10-20; First posted 2017-11-17 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2019-12

CONDITIONS: Hematopoietic Cell Transplant

STUDY DESIGN:
Intervention Model Description: interactive group drumming sessions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interactive group drumming sessions (Experimental): Participants will be involved in four interactive group drumming sessions (10-30 minutes each) and complete surveys and questionnaires about music and quality of life.
  Interventions: Behavioral: interactive group drumming sessions

INTERVENTIONS:
Behavioral: interactive group drumming sessions — interactive group drumming sessions

SUMMARY:
The purpose of this research is to determine if it is possible to perform group drumming as an intervention during HCT, to begin to understand how interactive group drumming during HCT treatment affects patients' well-being (good and bad) during the treatment course and in the first four weeks after completion of the drumming sessions.

DETAILED DESCRIPTION:
The purpose of this research is to determine if it is possible to perform group drumming as an intervention during HCT, to begin to understand how interactive group drumming during HCT treatment affects patients' well-being (good and bad) during the treatment course and in the first four weeks after completion of the drumming sessions.

ELIGIBILITY:
Inclusion Criteria:

* People who are at least 18 years old and are scheduled for HCT
* Individuals must be able to understand and willing to sign a written informed consent form

Exclusion Criteria:

* People who are too ill to participate, i.e., while they are in contact isolation or have low platelets (less than 20,000/mcl) will not participate until their condition has improved.
* Patients receiving outpatient HCT except patients with multiple myeloma. Patients with multiple myeloma may participate in the study even though they tend to spend nights away from the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Rate of participation | Up to 1 week after hematopoietic cell transplant (HCT)
  Defined as the number of subjects willing to participate in the interactive group drumming (IGD) divided by the number approached and asked to participate. These rates will be reported, along with the corresponding 95% confidence interval.
Rate of completion | Up to 1 week after HCT
  Defined as the ratio of (the number of individuals who successfully complete the study [4 sessions of IGD (about 20 minutes [min.] each)], with two pre-and post- surveys [8 minutes total, and two questionnaires (10 minutes total) about 160 minutes total time]) relative to the number of individuals who consent to the study (the number from the numerator of the first ratio [participation]). These rates will be reported, along with the corresponding 95% confidence interval.

SECONDARY OUTCOMES:
Gather patient-reported data to suggest how participants respond to interactive group drumming (IGD) | Baseline up to 4 weeks after completion of IGD
  Will be assessed by STADID Short Form Y-1. The after-IGD session measure will include a patient satisfaction item as well. The mean and standard deviation for each of these measures will be calculated.
Determine optimum length of session | Up to 4 weeks after completion of IGD
  Will be assessed by comparing actual length of session reported on facilitator post-session observation forms with participant satisfaction as reported in post-session. The mean and standard deviation for each of these measures will be calculated.
Gather patient-reported information to study whether the effect of interactive group drumming (IGD) on targeted variables is more pronounced in successive sessions | Baseline up to 4 weeks after completion of IGD
  Targeted variables defined as anxiety, energy mood, distress, relaxation, pain, and patient satisfaction. Will compare for each participant. The mean and standard deviation for each of these measures will be calculated.
Effect of support care provider (SCP) presence for each participant and among participants | Up to 4 weeks after completion of IGD
  Will use a non-parametric test to compare difference in item scores with and without SCP presence.
Change in physiological response to interactive group drumming (IGD) | Baseline up to 1 week after HCT
  Will be calculated at three time points during the session; repeated measures analysis of variance will be used to detect changes over the 3 readings.
Gather patient-reported information to suggest the optimal number of interactive group drumming (IGD) sessions | Baseline up to 4 weeks after completion of IGD
  Will be assessed by STADID Short Form Y-1. The after-IGD session measure will include a patient satisfaction item as well. The mean and standard deviation for each of these measures will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Richard McQuellon, PhD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT03345433/ICF_000.pdf